CLINICAL TRIAL: NCT05091333
Title: FASENRA Regulatory Postmarketing Surveillance in Korea
Acronym: FASENRA rPMS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00043
Record Dates: First submitted 2021-09-30; First posted 2021-10-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Asthma, EGPA(Eosinophilic Granulomatosis With Polyangiitis)
MeSH Terms: conditions — Asthma; Churg-Strauss Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
As part of a post approval commitment, the MFDS has requested a study to characterize safety in patients who are treated with FASENRA for severe eosinophilic asthma and/or eosinophilic granulomatosis with polyangiitis (EGPA) by physicians in normal clinical practice settings. This study is designed to confirm or assess the known safety profile or identify previously unsuspected adverse reactions and to evaluate the effectiveness of FASENRA under conditions of routine daily medical practice in Korea.

DETAILED DESCRIPTION:
This is a local, prospective, non-interventional, observational study is designed to evaluate safety and effectiveness of FASENRA in real world clinical practice setting in Korea. Adult patients with severe eosinophilic asthma and/or eosinophilic granulomatosis with polyangiitis (EGPA) who are initiating FASENRA for the first time as indicated by the MFDS will be included. At least 45 patients are followed for up 24 weeks and/or 48 weeks.

Patients will be treated as part of routine practice at Korean healthcare centers by accredited physicians. Each investigator will sequentially enroll patients who are initiating FASENRA for the first time and receive at least one dose until the target number of patients per center is reached. The characteristics of the study population and the FASENRA treatment schedule should be consistent with those described in the local product information at the time of enrolment (as the local product information may change). The study will enrol patients until the target number is reached.

All patients will be evaluated for safety during FASENRA use or for 30 days after their last dose of the surveillance drug if patients discontinued FASENRA before 24 weeks. Investigator's follow up of adverse events can be conducted by mail, phone calls, or e-mail for patients who discontinue early. The decision about the duration and discontinuation of treatment is solely at the discretion of the treating investigator with agreement of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years and older
2. Patients with severe asthma with an eosinophilic phenotype eligible for first time treatment with FASENRA according to the indication as indicated in the locally approved prescribing information
3. Patients with evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. Hypersensitivity to the active substances or to any of the excipients
2. Current participation in any interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older, Patients with severe asthma with an eosinophilic phenotype eligible for first time treatment with FASENRA according to the indication as indicated in the locally approved prescribing information
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Percentage (%) of AEs and SAEs in patients who are treated with FASENRA | 24 or 48 weeks
Nature (type) of AEs in patients who are treated with FASENRA | 24 or 48 weeks
Incidence of AEs in patients who are treated with FASENRA | 24 or 48 weeks
Severity of AEs in patients who are treated with FASENRA | 24 or 48 weeks
Nature of unexpected adverse drug reactions in patients who are treated with FASENRA | 24 or 48 weeks
Incidence of unexpected adverse drug reactions in patients who are treated with FASENRA | 24 or 48 weeks
Severity of unexpected adverse drug reactions in patients who are treated with FASENRA | 24 or 48 weeks

SECONDARY OUTCOMES:
Number of exacerbation | 24 or 48 weeks
Numbers of hospitalizations or ER visits due to asthma exacerbation | 24 or 48 weeks
Overall investigator's assessment on the outcome of the treatment: "Well control", "Partly control", "Uncontrolled" | 24 or 48 weeks
Overall investigator's assessment on any of the criteria below | 24 or 48 weeks
  EGPA Remission (defined as BVAS = 0 and prednisolone/prednisone dose ≤ 4 mg/day)
  ≥ 50% reduction in average daily prednisolone/prednisone dose EGPA relapse free during treatment period

OTHER OUTCOMES:
Pre-bronchodilator FEV1(mL), if available | 24 or 48 weeks
Peripheral blood eosinophil count, if available | 24 or 48 weeks
FeNO, if available | 24 or 48 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Research Site, Busan
  - Research Site, Gangneung-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Ulsan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250R00043&attachmentIdentifier=2f1a0742-aeaf-4b4e-8e61-b70eff34de22&fileName=D43250R00043_Redacted_CSR_Synopsis.pdf&versionIdentifier=